CLINICAL TRIAL: NCT02689921
Title: A Phase II Study of NEOADjuvant Aromatase Inhibitor and Pertuzumab/Trastuzumab (NEOADAPT)
Brief Title: NEOADjuvant Aromatase Inhibitor and Pertuzumab/Trastuzumab for Women With Breast Cancer
Acronym: NEOADAPT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Ahn, Principal Investigator, Midwestern Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MZ2016006; ML30001 (Other: Genentech, Inc.)
Record Dates: First submitted 2016-02-04; First posted 2016-02-24 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Letrozole; Anastrozole; Leuprolide; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Biological Therapy (Experimental): Subjects will receive an aromatase inhibitor for the duration of the study [exemestane (tablet, oral, 25 mg/day), letrozole (tablet, oral, 2.5 mg/day) or anastrozole (tablet, oral, 1 mg/day)]. Premenopausal subjects will receive leuprolide acetate (11.25 mg, intramuscular injection, 3-month intervals).
  Pertuzumab will be given by intravenous infusion in 3-week cycles until disease progression (Cycle 1 Day 0: 840 mg, infused over 60-90 minutes; subsequent cycles: 420 mg, infused over 30-60 minutes).
  Trastuzumab will be given by intravenous infusion in 3-week cycles until disease progression (Cycle 1 Day 0: 8 mg/kg, infused over 60-90 minutes; subsequent cycles: 6 mg/kg, infused over 30-60 minutes)
  Interventions: Drug: Exemestane; Drug: Letrozole; Drug: Anastrozole; Drug: Leuprolide Acetate; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Exemestane — Aromatase inhibitor
  Other Names: Aromasin
Drug: Letrozole — Aromatase inhibitor
  Other Names: Femara
Drug: Anastrozole — Aromatase inhibitor
  Other Names: Arimidex
Drug: Leuprolide Acetate — Luteinizing Hormone-Releasing Hormone agonist
  Other Names: Lupron; Lupron Depot
Drug: Pertuzumab — Monoclonal antibody (HER2/neu receptor antagonist)
  Other Names: Perjeta
Drug: Trastuzumab — Monoclonal antibody (HER2/neu receptor antagonist)
  Other Names: Herceptin

SUMMARY:
This is a prospective, single-arm, phase II study of 32 evaluable patients treated with NEOADjuvant Aromatase inhibitor and Pertuzumab/Trastuzumab (NEOADAPT) without chemotherapy for hormone receptor positive (HR+), [i.e. Estrogen Receptor positive (ER+) and/or Progesterone Receptor positive (PR+)] HER2+ localized, non-metastatic stage I - IIb breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide signed, written informed consent
* Histologically or cytologically confirmed non-metastatic adenocarcinoma of the breast (stage I-II)
* Candidate for curative-intent treatment
* ER+ and/or PR+ and HER2-positive (Fluorescence In Situ Hybridization-positive or 3+ by Immunohistochemistry staining)
* Life expectancy greater than 5 years
* Left Ventricular Ejection Fraction > 50% at baseline (within 30 days of day 0)
* Eastern Cooperative Oncology Group performance status ≤2
* Absolute Neutrophil Count >1000/µL
* Platelets ≥50,000/µL
* Hemoglobin >8.0 g/dL,
* Creatinine ≤3.0 x upper limit of normal (ULN)
* Bilirubin ≤3.0 x ULN
* Aspartate aminotransferase or Alanine aminotransferase <5.0 x ULN
* Negative serum pregnancy test for women <12 months after the onset of menopause unless surgically sterilized
* Agreement by women of childbearing potential and male participants with partners of childbearing potential to use a "highly effective", non-hormonal form of contraception or two "effective" forms of non-hormonal contraception by the patient and/or partner.

Exclusion Criteria:

* Active infection
* Presence of known metastases (stage IV disease)
* Pregnant or lactating women
* Prior chemotherapy or radiation therapy for the primary breast cancer
* Concomitant malignancies or previous malignancies within the last 5 years except adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* History of significant cardiac disease, cardiac risk factors or uncontrolled arrhythmias
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary or metabolic disease including diabetes, wound healing disorders, ulcers or bone fractures)
* Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start or anticipated need for major surgery during the course of study treatment
* Current known infection with Human Immunodeficiency Virus (HIV), Hepatitis B virus (HBV) or Hepatitis C Virus (HCV)
* Receipt of intravenous antibiotics for infection within 14 days prior to receiving study treatment
* Current chronic daily treatment with corticosteroids (dose >10 mg/day methylprednisolone equivalent) except inhaled steroids
* Known hypersensitivity to any of the study drugs
* Assessment by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of Pathological Response | One year
  The presence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy. Pathological complete response (pCR) is defined as the absence of residual invasive cancer.

SECONDARY OUTCOMES:
Duration of Treatment | One year
  Median number of days between Day 0 (first treatment of trastuzumab and pertuzumab) and three weeks after the last dose of neoadjuvant trastuzumab and pertuzumab on treatment protocol.
Evidence of Radiographic Response | Assessed every 12 weeks up to one year
  Change in dimensions (millimeters) of target lesions (along long axis) and non-target lesions (along long axis for non-lymphatic lesions and short axis for lymph nodes) as observed by Magnetic Resonance Imaging and quantified by modified RECIST 1.1 criteria.
Measurement of Left Ventricular Ejection Fraction (LVEF) | Assessed every 12 weeks up to one year
  Determination of cardiac function as measured by echocardiogram or multi-gated acquisition scan (MUGA).
Mammaprint Genomic Analysis | One year or up to 3 months after definitive surgery
  Mammaprint will estimate the risk level of the subject's tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Ahn, MD, Principal Investigator — Midwestern Regional Medical Center
Locations (2):
- United States (2):
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Cancer Treatment Centers of America at Midwestern Regional Medical Center, Zion, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT02689921/Prot_SAP_000.pdf